CLINICAL TRIAL: NCT05192343
Title: Effects of Virtual Reality and Nature Sounds on Pain and Anxiety During Hysterosalpingography: Randomized Controlled Study
Brief Title: Effects of Virtual Reality and Nature Sounds on Pain and Anxiety During Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sümeyye BAL (Other)
Responsible Party: Sponsor-Investigator, Sümeyye BAL, Lecturer Dr., Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/435
Record Dates: First submitted 2022-01-12; First posted 2022-01-14 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Women's Health

STUDY DESIGN:
Intervention Model Description: This randomized controlled study was conducted at Ondokuz Mayis University Training and Research Hospital, Obstetrics and Gynecology polyclinic between February 2022 and August 2022. The CONSORT (Consolidated Standards of Reporting Trials) guidelines for reporting randomised controlled trials (RCTs) has been used to describe the methods.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality and nature sounds (Experimental): After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and visual analogue scale scoring scale for pain will apply to both groups by face to face interview during the day giving appointment for hysterosalpingography. Immediately after the questionnaires will apply, before and during the HSG procedure, the Virtual Reality and nature sounds application group watch a video with a nature view with virtual reality glasses.Glasses will introduce before the procedure. Before the procedure started, glasses will put on and training will given to continue watching the video by wearing glasses during the procedure. The women will be included in the Virtual Reality and nature sounds intervention group will make to watch a video with a nature view for 15 minutes and listening nature sounds before and during the HSG procedure. Each woman was shown the same video.
  Interventions: Device: Virtual Reality and nature sounds
- nature sounds (Experimental): After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and visual analogue scale scoring scale for pain will apply to both groups by face to face interview during the day giving appointment for hysterosalpingography. Immediately after the questionnaires will apply, a nature-based sound will play to the women in the nature sounds group before and during the HSG shooting.Listening to nature-based sound will perform for a total of 15 minutes half an hour before the HSG procedure, and for 15 minutes during the procedure, for a total of 30 minutes.
  Interventions: Other: nature sounds
- control group (No Intervention): Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention will perform. Both groups will re-evaluated using the same scales after the hysterosalpingography.

INTERVENTIONS:
Device: Virtual Reality and nature sounds — After obtaining informed consent, the data collection form, Spielberger State Anxiety Scale and VAS scoring scale for pain were applied to both groups by face to face interview during the day giving appointment for HSG. Before and during the HSG shooting, the virtual reality and nature sounds application group watched a video with a nature view with virtual reality glasses and listening nature sounds.
  Glasses were introduced before the procedure. Before the procedure started, glasses were put on and training was given to continue watching the video by wearing glasses during the procedure.
  The women include in the virtual reality and nature sounds application group will make to watch a video with a nature view with nature sounds for 15 minutes before and during the HSG procedure.
  Each woman was shown the same video.
  Arms: Virtual Reality and nature sounds
Other: nature sounds — After obtaining informed consent, the data collection form, Spielberger State Anxiety Scale and VAS scoring scale for pain were applied to both groups by face to face interview during the day giving appointment for HSG. Before the procedure started, glasses will put on and training was given to continue. After the groups were formed, a nature-based sound was played to the women in the nature sounds group before and during the HSG shooting.
  Listening to nature-based sound will perform for a total of 15 minutes half an hour before the HSG procedure, and for 15 minutes during the procedure, for a total of 30 minutes.
  Arms: nature sounds

SUMMARY:
The aim of this study is to demonstrate the effects of virtual reality and nature sounds on pain and anxiety during hysterosalpingography.

DETAILED DESCRIPTION:
Infertility treatment is a stressful and anxious process that begins when couples are diagnosed with infertility. Although this process may seem like a simple medical intervention, the treatment stages affect the couple in many ways when it is deepened. Infertility treatment is a process that requires the active participation of couples against emotional and physical difficulties. The treatment process is a period in which couples should be in constant communication with healthcare professionals, as well as intensive routine and surgical procedures.In this process, medical and surgical treatment methods are used. In the literature, it is stated that 85-90% of the problems that cause infertility are solved with medical and surgical treatment. In the evaluation of infertile couples, hysterosalpingography (HSG) is a invasive radiologic procedure to visualize uterine cavity and tubes after contrast enhancement. HSG plays an important diagnostic role in finding the cause of infertility and in deciding the line of management.The aim of this study is to demonstrate the effects of virtual reality and nature sounds on pain and anxiety during hysterosalpingography. This randomized controlled study will conduct at Ondokuz Mayıs University Training and Research Hospital, Obstetrics and Gynecology polyclinic between February 2022 and August 2022. Volunteer women undergoing HSG as part of infertility evaluation will be includ. Participants will randomly assigned to the Virtual Reality and nature sounds intervention, nature sounds intervention or the control group using a computer-generated list. A data collection form including socio-demographic and obstetric characteristics such as age, educational status, place to live, duration of infertility, previous pregnancies, births, abortion/curettage numbers, Spielberger State Anxiety Scale and Visual Analog Scale for pain and Visual Analog Scales for satisfaction will use for each patient. After obtaining written informed consent, the data collection form, Spielberger State Anxiety Scale and VAS pain scoring scale will be applied to both groups by face to face interview during the day giving appointment for HSG. Immediately after the questionnaires were applied, the nurse gave virtual reality glasses and headphone to intervention group for before HSG and while HSG totally 30 minutes. The nurse gave to nature sounds intervention group headphone. After the groups will formed, a nature-based sound will listen to the women in the nature sounds group before and during the HSG procedure. Listening to nature-based sound will perform for a total of 15 minutes half an hour before the HSG procedure, and for 15 minutes during the procedure, for a total of 30 minutes. Participants in the control group received standard care (verbal information about procedure and a short written information about the procedure) and no intervention (nature sounds or virtual reality) will perform.The IBM SPSS (Statistical package for the Social Sciences) 23.0 package program will use to evaluate the data obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

* Wanting to participate in the study,
* being literate,
* over 18 years,
* at least primary school graduate,
* without a diagnosed psychiatric illness,
* not have mental insufficiency and communication problems,
* have no hearing problems,
* without drug sensitivity and allergy,

Exclusion Criteria:

* illiterate,
* with a diagnosed psychiatric illness,
* mental deficiency and communication problems,
* under 18 years old,
* who did not want to participate in the research,
* having hearing problems
* drug sensitivity and allergy,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Spielberger State Anxiety Scale | 30 minutes
  The inventory was developed by Spielberger, Gorsuch, and Lushene in 1970. An adaptation, validity, and reliability study of the State-Trait Anxiety Scale in Turkish was conducted by Oner and Le Compte in 1983. The scale consists of two subdimensions: the state anxiety has 20 items and is used to determine what is felt at a specific moment under certain conditions, and the trait anxiety has 20 items and is used to determine what has been felt in the last 7 days. High scores from each subscale indicate a high level of anxiety. The Cronbach's a for the STAI ranges from 0.83 to 0.87
Visual Analog Scale For Satisfaction | 10 minutes
  Visual Analog Scale Satisfaction level was measured using the visual analog scale (VAS). VAS is used to convert some numerically unmeasured values to numeric values. VAS is a continuous scale that comprises a horizontal line or a vertical line, usually 10 cm (100 mm) in length. On one end of the scale is the statement, "I am not satisfied at all" (zero points), whereas the statement at the other end is "very satisfied." Patients were asked to mark their satisfaction levels on this scale of 100 mm.
Visual Analog Scale for pain | 10 minutes
  The pain was assessed using 0-100 mm VAS for determining perceptions of pain during the procedure. This scale is widely used and has demonstrated reliability and validity in the measurement of acute pain. A high score on the scale indicated a high level of pain and a score of 0 pointed to no pain at all (Bijur, Silver, & Gallagher, 2001). Each participant was asked to mark her current level of perceived pain along the scale, with the number corresponding to the marked point recorded as the pain score

CONTACTS AND LOCATIONS:
Overall Officials: Emine KOÇ, Asst.Prof, Study Chair — Ondokuz Mayıs University; Nazlı BALTACI, Asst.Prof, Study Director — Ondokuz Mayıs University; Elif KETEN EDİS, Lecturer, Study Chair — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Atakum, Turkey (Türkiye)

REFERENCES:
- [Background] Agwu, K. K., & Okoye, I. J. (2007). The effect of music on the anxiety levels of patients undergoing hysterosalpingography. Radiography, 13(2), 122-125.